CLINICAL TRIAL: NCT03371667
Title: A Multi-center Randomized in Double-blinded Phase III Study Comparing Standard Care Therapy Alone Versus Corticosteroids and Low-dose Methotrexate (MTX) for the First-line Treatment of Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Brief Title: To Compare the Efficacy of the Addition of Methotrexate (MTX) to Current Standard Acute Graft-versus-host Disease (GVHD) First-line Treatment With Corticosteroids
Acronym: MTX-aGVHD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-K 16-150; 2017-002691-98 (EudraCT Number)
Record Dates: First submitted 2017-07-31; First posted 2017-12-13 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Allogeneic Disease; GVH - Graft Versus Host Reaction; GVHD, Acute; Stem Cell Transplant Complications
Keywords: Hematopoietic Stem Cell; Methotrexate; Corticosteroids therapy; Acute GVHD; Allogenic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): * 5mg/Kg/day methotrexate for 4 weeks then 3 mg/m2 every two weeks for 12 weeks
  * 2mg/kg/day PO prednisone prednisone (or 1.6 mg/kg/day IV methylprednisolone) once daily.
  * 10 mg po or iv lederfolin after each MTX administration
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): * Once a week placebo for 4 weeks then every two weeks for 12 weeks
  * 2 mg/kg/day PO prednisone (or 1.6 mg/kg/day IV methylprednisolone) once daily.
  * 10 mg po or iv lederfolin after each placebo administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 5 mg/m2 will be given once week for 4 weeks, then 3 mg/m2 every two weeks for 12 weeks. Body surface area will be capped at 2 m2.
  Methotrexate will be given as an IV infusion over 15 minutes. All patients will received prednisone 2 mg/kg.day PO (or methylprednisolone 1.6 mg/Kg/day) for 3 days.
  For responding patients between day 4 and 28, the dose of prednisone must be at least 0.25 mg/kg/day prednisone (or 0.2 mg/kg/day methylprednisolone).
  All patients should receive a folinic acid supplementation 24 hours after each MTX/placebo administration.
  Lederfoldin 10 mg po or iv will be administered on days 2, 9, 16 and 23. Lederfoldin 10 mg po or iv will be administered on days 37, 51, 65, 79, 93 and 103.
  Arms: Methotrexate
Drug: Placebo — Placebo 5 mg/m2 will be given once week for 4 weeks, then 3 mg/m2 every two weeks for 12 weeks. Body surface area will be capped at 2 m2.
  Placebo will be given as an IV infusion over 15 minutes. All patients will received prednisone 2 mg/kg.day PO (or methylprednisolone 1.6 mg/Kg/day) for 3 days.
  For responding patients between day 4 and 28, the dose of prednisone must be at least 0.25 mg/kg/day prednisone (or 0.2 mg/kg/day methylprednisolone).
  All patients should receive a folinic acid supplementation 24 hours after each MTX/placebo administration.
  Lederfoldin 10 mg po or iv will be administered on days 2, 9, 16 and 23. Lederfoldin 10 mg po or iv will be administered on days 37, 51, 65, 79, 93 and 103.
  Arms: Placebo

SUMMARY:
Phase III randomized double-blinded trial designed to compare the efficacy of the addition of MTX to current standard acute GVHD first-line treatment with corticosteroids. The protocol will use a novel endpoint for benchmarking interventions based on a composite primary endpoint of GVHD-free and corticosteroids-free survival.

The primary endpoint of the trial will be the assessment of a composite endpoint of graft-versus-host disease-free and corticosteroids-free survival at 12 months after randomization

DETAILED DESCRIPTION:
This is a phase III randomized, multicenter, double blinded controlled study. Patients who develop clinically meaningful acute GVHD and who meet all other entry criteria will be randomized 1:1 to receive either corticosteroids and placebo ("standard of care", control arm) or the combination of low-dose MTX with corticosteroids as first-line therapy for acute GVHD (MTX; "experimental arm").

The primary analysis of this hypothesis generation study is to estimate the composite endpoint of GVHD-free and corticosteroids-free survival at 12 months after randomization in both treatment arms. In fact, it is more and more established that such composite endpoint is a clinically very relevant one because it represents ideal recovery from allo-SCT (Stem Cell transplantation) (at 1 year after acute GVHD diagnosis) and a measure of cure without ongoing morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (>=18 years old) with hematological diseases, who develop a first episode of acute GVHD (grade II-IV) requiring systemic therapy
* First allo-SCT, with any type of donor, stem cell source, GVHD prophylaxis or conditioning regimen
* Biopsy of acute GVHD target organ is recommended, but not required. Enrollment should not be delayed awaiting biopsy or pathology results
* The patient must have received no previous systemic immune suppressive therapy for treatment of acute GVHD, except for a maximum 72 hours of prior corticosteroid therapy
* Absolute neutrophil count (ANC) greater than 0.5 G/L
* Platelets count greater than 20 G/L
* Signed informed consent
* Affiliation to a social security system (recipient or assign)
* Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception until 6 months after the end of treatment.

Men with a partner of childbearing potential must agree to use a medically acceptable method of contraception until 6 months after the end of treatment.

Exclusion Criteria:

* Hyper-acute GVHD as defined by the MD Anderson's criteria (Saliba, de Lima et al. 2007)
* Flare of GVHD in a patient already on corticosteroid treatment
* Overlap chronic GVHD as defined by the NIH Consensus Criteria (Jagasia, Greinix et al. 2015)
* MTX given within 7 days of enrollment
* Active uncontrolled infection
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal
* Acute GVHD after donor lymphocytes infusion (DLI)
* Other systemic drugs for GVHD treatment (including extra-corporeal photopheresis)
* If any prior steroid therapy (for indication other than GVHD), treatment at doses > 0.5 mg/kg/day methyl-prednisolone within 7 days prior to onset of acute GVHD
* Patients who are pregnant, breast feeding, or if sexually active, unwilling to use effective birth control for the duration of the study
* Patient on dialysis
* Patients with veno-occlusive disease of the liver or with significant liver abnormalities who in the judgment of the treating physician cannot receive MTX
* Patients requiring after inclusion in the protocol the continuation of one or more of the following medication: probenecide, trimethoprime (alone or in combination with sulfametoxazole), phenylbutazone or yellow fever vaccine
* Patients with a history of intolerance/allergy to MTX
* Hypersensitivity to the active substance or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization. | Evaluation will be performed at time of inclusion
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (1). | Evaluation will be performed before start of MTX at the randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (2). | Evaluation will be performed at Day 8
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (3). | Evaluation will be performed at Day 15
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (4). | Evaluation will be performed at Day 22
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (5). | Evaluation will be performed at Day 28
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (6). | Evaluation will be performed at Day 36
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (7). | Evaluation will be performed at Day 50
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (8). | Evaluation will be performed at Day 56
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (9). | Evaluation will be performed at Day 64
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (10) | Evaluation will be performed at Day 78
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (11). | Evaluation will be performed at Day 92
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (12). | Evaluation will be performed at Day 102
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (13). | Evaluation will be performed at 5 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (14). | Evaluation will be performed at 6 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (17). | Evaluation will be performed at 9 months after randomization .
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of graft-versus-host disease-free at 12 months after randomization (18). | Evaluation will be performed at 12 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (19). | Evaluation will be performed at time of inclusion.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (20). | Evaluation will be performed before start of MTX at the randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (21). | Evaluation will be performed at Day 8.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (20). | Evaluation will be performed at Day 15.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (21). | Evaluation will be performed at Day 22.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (22). | Evaluation will be performed at Day 28.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (23). | Evaluation will be performed at Day 36
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (24). | Evaluation will be performed at Day 50.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (25). | Evaluation will be performed at Day 56.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (26). | Evaluation will be performed at Day 64.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (27). | Evaluation will be performed at Day 78.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (28). | Evaluation will be performed at D92.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (29). | Evaluation will be performed at Day 102.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (30). | Evaluation will be performed at 5 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (31). | Evaluation will be performed at 6 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (32). | Evaluation will be performed at 9 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.
Assessment of a composite endpoint of corticosteroids-free survival at 12 months after randomization (33). | Evaluation will be performed at 12 months after randomization.
  GVHD-free survival is defined as absence of initiation of additional GVHD therapy or development of chronic GVHD requiring systemic therapy, and corticosteroids-free survival as absence of continuation of corticosteroids above a dose of 0.15 mg/Kg day.

SECONDARY OUTCOMES:
The incidence of severe adverse events within the first 12 months after randomization | 12 months after randomization
The proportion of complete remission (CR), very good partial response (VGPR), partial response (PR), mixed response (MR), no response (NR) and progression at day 28, day 56 and best response within the first 12 months after randomization. | at day 28, day 56 and best response within the first 12 months after randomization.
The proportion of GVHD flare within the first 12 months after randomization. | 12 months after randomization
Cumulative incidence of overall and severe chronic GVHD as assessed by NIH Consensus Criteria within the first 12 months after randomization(Jagasia, Greinix et al. 2015, Lee, Wolff et al. 2015). | within the first 12 months after randomization
Incidence of systemic of infection and CMV(cytomegalovirus ) reactivation within 3 months after randomization | within 3 months after randomization
Incidence of EBV (Epstein-Barr virus) reactivation and post-transplant lymphoproliferative disease within 12 months after randomization | within 12 months after randomization
Cumulative incidence of non-relapse mortality within the first 12 months after randomization. | 12 months after randomization
Corticosteroids-free, disease-free and overall survival within the first 12 months after randomization. | 12 months after randomization
Immune recovery and microbiota: number of patients with complete immune recovery (lymphocytes and dendritic cells) and correction of microbiota dysbiosis within the first 12 months | 12 months after randomization
Quality of Life (QoL)-1 | 12 Months
  Evaluation by 1 questionnaire: EORTC QLQ-C30 (quality of life questionnaire) (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30)
Quality of Life (QoL)-2 | 12 Months
  Evaluation by 1 questionnaire: FACT-BMT (Functional Assessment of Cancer Therapy - Bone Marrow Transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital - Hematology Department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided